CLINICAL TRIAL: NCT04966052
Title: Effect of COPD Co-infection With Tuberculosis on Th17 Cell Differentiation and Its Significance
Brief Title: COPD Co-infection With Tuberculosis on Th17 Cell Differentiation
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Geriatric Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2017390
Record Dates: First submitted 2021-07-04; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2020-07

CONDITIONS: Tuberculosis Infection; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Latent Tuberculosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The distribution of T-cell subtypes, including CD4+ and CD8+ T cells and Th17 cells, in blood specimens and alveolar lavage fluid was detected by flow cytometry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COPD combined with TB group: COPD combined with pulmonary TB infection
  Interventions: Other: No intervention
- COPD non-TB control group: COPD combined without pulmonary TB infection
- TB non-COPD control group: pulmonary TB infection without COPD
- Non-smoking non-TB control group: Non-smoking without pulmonary TB infection

INTERVENTIONS:
Other: No intervention — No intervention
  Groups: COPD combined with TB group

SUMMARY:
This project will observe and follow up the changes of pulmonary function and CT in patients with smoking combined with pulmonary tuberculosis, and measure the ratio of Th1 cells, Th17 cells, macrophages and neutrophils and the secretion of factors such as TNF-α, IFN-γ and IL-17 in pulmonary blood and alveolar lavage fluid.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) and tuberculosis are major global health problems, and acquired and acquired immunity play an important role in COPD and tuberculosis, and there is an interaction between COPD and tuberculosis, but the exact mechanism is not clear. Pre-existing TB infection is an independent risk factor for COPD and can aggravate pulmonary function and increase hospitalization and mortality in COPD patients. In COPD patients, Th1 and Th17 cells are involved in the development of COPD and emphysema through activation of macrophages and recruitment of neutrophils, while matrix metalloproteinases (MMPs) of macrophage and neutrophil origin are involved in the formation of tuberculosis cavities, and cytokines such as TNF-α, IFN-γ, IL-17 are involved in the mechanism of their destruction, IL-17 restricts the expression of HIF-1α to inhibit the development of TB granulomas, and CT analysis revealed that combined TB exacerbates emphysema in COPD patients. The above evidence suggests that tuberculosis plays an important role in the formation of emphysema in COPD. In this project, we will observe and follow up the changes of pulmonary function and CT in patients with smoking combined with pulmonary tuberculosis, and examine the ratio of Th1 cells, Th17 cells, macrophages and neutrophils and the secretion of TNF-α, IFN-γ, and IL-17 in pulmonary blood and alveolar lavage fluid.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* age ≧ 40

Exclusion Criteria:

* Presence of other chronic respiratory diseases other than COPD, such as asthma, bronchiectasis, interstitial lung disease, etc.
* History of chest and lung surgery.
* History of malignancy.
* Autoimmune disease.
* Long-term oral glucocorticoids, immunosuppressants and inhaled glucocorticoids.
* Mental abnormalities, cognitive impairment, inability to cooperate with pulmonary function and other tests.
* Acute stage of infection, such as lung infection, urinary tract infection and gastrointestinal tract infection, etc.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients seen at Peking University Third Hospital and Beijing Geriatric Hospital Respiratory Department from April 1, 2018 to April 1, 2020
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Differentiation of Th17 cells | Day 1
  Distribution of T cell subtypes, including CD4+, CD8+ T cells and Th17 cells, in blood specimens and alveolar lavage fluid by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Sun, MD, Principal Investigator — Peking University 3rd Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gai X, Cao W, Rao Y, Zeng L, Xu W, Wu H, Li G, Sun Y. Risk factors and biomarkers for post-tuberculosis lung damage in a Chinese cohort of male smokers and non-smokers: protocol for a prospective observational study. BMJ Open. 2023 Oct 9;13(10):e065990. doi: 10.1136/bmjopen-2022-065990. PMID 37813532